CLINICAL TRIAL: NCT04398290
Title: Randomized Controlled Trial Of A Delivered Continuously By Nasal Cannula For The Treatment Of Patients With COVID-19 And Mild To Moderate Hypoxemia Requiring Supplemental Oxygen
Brief Title: iNOPulse for COVID-19
Acronym: NO-COVER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB AND FDA REVIEWS DEFERRED
Sponsor: Roger Alvarez (Other)
Collaborators: Bellerophon Therapeutics (Unknown)
Responsible Party: Sponsor-Investigator, Roger Alvarez, Assistant Professor of Clinical Medicine Pulmonary Vascular Diseases, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200449
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Hypoxemia; Hypoxemic Respiratory Failure
Keywords: hypoxemia; respiratory failure; COVID-19; inhaled nitric oxide
MeSH Terms: conditions — COVID-19; Hypoxia; Respiratory Insufficiency | interventions — Nitrogen; nitrox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iNOpulse Treatment Group (Experimental): Participants in this group will receive iNO delivered continuously together with supplemental oxygen by nasal cannula during hospitalization for up to 28 days.
  Interventions: Drug: Inhaled nitric oxide (iNO); Drug: Oxygen gas
- Placebo Group (Active Comparator): Participants in this group will receive nitrogen gas delivered continuously together with supplemental oxygen by nasal cannula during hospitalization for up to 28 days
  Interventions: Drug: Nitrogen gas; Drug: Oxygen gas

INTERVENTIONS:
Drug: Inhaled nitric oxide (iNO) — iNO Pulse 250 mcg/kg ideal body weight (IBW)/hour
  Arms: iNOpulse Treatment Group
Drug: Nitrogen gas — 250 mcg/kg ideal body weight (IBW)/hour
  Arms: Placebo Group
Drug: Oxygen gas — Supplemental oxygen administered via nasal cannula

SUMMARY:
This randomized, controlled trial will assess the efficacy and safety of pulsed iNO in subjects with COVID-19 who are hospitalized and require supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Proven COVID-19 viral infection. Non-confirmed highly suspicious suspects may be enrolled.
3. Presence of radiographic findings compatible with pneumonia/pneumonitis.
4. Patients requiring at least 3 L/m oxygen via nasal canula to maintain O2 above 92%.
5. Female subjects of childbearing potential must have a negative pre-treatment pregnancy test (serum or urine).
6. Willing and able to comply with treatment schedule and study procedures.

Exclusion Criteria:

1. Patient with severe hypoxemia who are unable to maintain an oxygen saturation (SpO2) > 88% on a maximum supplemental oxygen of 6 L/m by nasal cannula and a non-rebreather facemask.
2. Participating in any other clinical trial for COVID-19
3. Pregnancy, or positive pregnancy test in a pre-dose examination.
4. Open tracheostomy.
5. Clinical contra-indication, as deemed by the PI or their designee.
6. Use of a nitric oxide donor agent such as nitroglycerin or drugs known to increase methemoglobin such as intravenous lidocaine, or topical benzocaine or dapsone at screening.
7. Known history or clinical evidence of heart failure or left ventricular dysfunction (LVEF < 45%).
8. Significant hemoptysis
9. Unable to provide informed consent (proxy consent is acceptable if available)
10. Any of the following conditions at time of possible enrollment: Fulminant Liver Failure, Acute Coronary Syndrome , Renal Failure requiring dialysis, Bacteremia, Shock, Cardiac arrest, Cardiac arrhythmia requiring acute treatment, Delirium / Encephalopathy, Severe Disseminated Intravascular Coagulation, Gastrointestinal hemorrhage, Hypoglycemia, Pneumothorax, Rhabdomyolysis / Myositis, Seizures, or Acute Stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Up to 14 days
  As assessed per treating physician's discretion.
Incidence of adverse events | Up to 6 hours
  Incidence of hypoxemia and hypotension as assessed per treating physician's discretion.
Incidence of methemoglobinemia | Up to 14 days
  Incidence of increase to > 5% total methemoglobin as assessed by pulse oximetry.

SECONDARY OUTCOMES:
Number of participants with progression of respiratory failure | Up to 14 days
  Worsening respiratory status as defined by any one of the following: Implementation of High Flow Nasal Cannula (HFNC), non-rebreather mask, non-invasive ventilation, intubation and mechanical ventilation or need for intubation (in the event the patient is not intubated due to do not intubate (DNI) or do not resuscitate (DNR) status).
Time until resolution of hypoxemia | Up to 14 days
  The number of days until hypoxemia is resolved as per treating physician assessment
Incidence of mortality | Up to 28 days
  Incidence of death during hospitalization and after discharge up to 28 days
Duration of hospitalization | Up to 28 days
  Number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Alvarez, D.O., Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospitals & Clinics, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No